CLINICAL TRIAL: NCT03166982
Title: Comparative Effectiveness Clinical Early of Transvaginal and Laparoscopic Approaches for Drainage of Tubo -Ovarian Abscess. Randomized Noninferiority
Brief Title: Drainage of Tubo - Ovarian Abscess: DTOA
Acronym: DTOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0283; 2016-A00961-50 (Other: 2016-A00961-50)
Record Dates: First submitted 2016-10-10; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2016-10

CONDITIONS: Tubo-ovarian Abscess
Keywords: Tubo-ovarian abscess; Transvaginal drainage; Laparoscopic treatment
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Intervention Model Description: Participants receive an intervention throughout the protocol
Masking Description: Open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopy (Experimental): the tubo-ovarian abscess should be drained by interventional radiology, preferably by transvaginal or laparoscopic
  Interventions: Procedure: laparoscopic approach
- ultrasound-guided puncture (Experimental): The transvaginal echo guided puncture to replace the first laparoscopy because of its less invasive nature, this is a simple act, fast, possible under mild sedation, the cost is still lower than laparoscopy
  Interventions: Procedure: transvaginal approach

INTERVENTIONS:
Procedure: transvaginal approach
  Arms: ultrasound-guided puncture
Procedure: laparoscopic approach
  Arms: laparoscopy

SUMMARY:
The treatment of the acute phase of the complicated abscess tubo-ovarian relies on antibiotics more or less associated with surgical management in case of visible abscess, poor clinical tolerance (sepsis) and resistance to medical treatment. The CNGOF recommended in 2012 that the tubo-ovarian abscess are not within one antibiotic, and should be drained by interventional radiology, preferably by transvaginal or laparoscopic.

Furthermore the efficiency of drainage by ultrasound puncture performed vaginally was demonstrated. This approach tends to replace the first laparoscopy because of its less invasive, fast, easy to access, more acceptable and less cost compared to laparoscopy. This approach is recommended by the French and English colleges.

In total, the surgery in case of ATO is necessary, it is always coupled with antibiotics. Several surgical approaches are possible, laparotomy, laparoscopy and ultrasound-guided puncture. No prospective comparative study has been done, for which we want to develop this study.

DETAILED DESCRIPTION:
Retrospective studies evaluating the efficacy of these two supported relate the same cure rates between the two techniques. According to the literature of Garbin O.and al in 2012, the success rate of transvaginal puncture is generally 93.6%. The largest series of Gjelland al in 2005 and covers 302 consecutive patients with ATO who underwent triple antibiotic therapy and transvaginal puncture, the success rate was 93.4%. The failures that required surgical management have frequently revealed endometriosis or cancer. To support laparoscopic, Raiga and al in 1996 studied the support of 36 retrospectively patients who underwent laparoscopic incisional and wash the abscess with a success rate of 100%. Moreover Reich and al in 1987 found 90% success on a review of 25 patients.

The transvaginal echo guided puncture to replace the first laparoscopy because of its less invasive nature, this is a simple act, fast, possible under mild sedation, the cost is still lower than laparoscopy. Some uncontrolled retrospective studies suggest that laparoscopy remains associated with prolongation of hospitalization time, it is also mentioned that the transvaginal puncture is better tolerated by the patient.

No study has compared these two techniques, which is why we propose this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a IGH with tubo-ovarian abscess visible on ultrasound or CT
* Ultrasound abscess> or equal to 2cm
* Abdominal pain syndrome
* Age 18 to 43 years
* understand french language
* No complicated: good hemodynamic tolerance, not broken
* These patients should be affiliated to the French Social Security and must have given informed participation agreement

Exclusion Criteria:

Patients with HIV (CD4 <200) or co-infections: immunosuppression

* Multi-Abdomen surgery
* Suspected malignant or borderline tumor
* Complicated abscess: rupture of the abscess, peritonitis, septic shock
* Postoperative pelvic abscess
* Patient minor
* During Pregnancy
* Patient having already been accounted for tubo-ovarian abscess in progress
* Not accessible abscess transvaginal puncture
* Patients unable major, patients suffering from mental pathology incompatible with informed consent, refusal to participate

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10-26 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical cure rate defined by a composite score as defined by O'Brien PC (Procedures for Comparing samples with multiple endpoints Biometrics 1984; 40: 1079-1087.) | at 72 hour
Clinical cure rate defined by a composite score as defined by O'Brien PC (Procedures for Comparing samples with multiple endpoints Biometrics 1984; 40: 1079-1087.) | at 1 month
Clinical improvement | at 72 hours and at 1 month
  apyrexia to 72 hours and 1 month and EVA to 72 hours and 1 month
Organic improvement | at 72 hours and at 1 month
  CRP Standards and GB to 72 hours and 1 month if initially high

SECONDARY OUTCOMES:
Duration of hospital stay | at day 0
Analgesia Type: general anesthesia versus sedation | at day 1
recurrent complications | at day 1
  Per Statement of complications and postoperative and rehospitalization
Operating Time | at day 1
Fertility prognosis by Mage score | at 3 months
prognosis of chronic pelvic pain score by adhesions at second look laparoscopy | at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie GREMEAU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Gjelland K, Ekerhovd E, Granberg S. Transvaginal ultrasound-guided aspiration for treatment of tubo-ovarian abscess: a study of 302 cases. Am J Obstet Gynecol. 2005 Oct;193(4):1323-30. doi: 10.1016/j.ajog.2005.06.019. PMID 16202721
- [Background] Granberg S, Gjelland K, Ekerhovd E. The management of pelvic abscess. Best Pract Res Clin Obstet Gynaecol. 2009 Oct;23(5):667-78. doi: 10.1016/j.bpobgyn.2009.01.010. Epub 2009 Feb 20. PMID 19230781
- [Background] Gerber B, Krause A. A study of second-look laparoscopy after acute salpingitis. Arch Gynecol Obstet. 1996;258(4):193-200. doi: 10.1007/s004040050123. PMID 8844136
- [Background] Le Bouedec G, Pouly JL, Canis M, Wattiez A, Abbas B, Mage G, Bruhat MA. [Acute salpingitis. Celioscopy before and after treatment: 110 cases]. J Gynecol Obstet Biol Reprod (Paris). 1991;20(5):680-4. French. PMID 1835469
- [Background] Raiga J, Canis M, Le Bouedec G, Glowaczower E, Pouly JL, Mage G, Bruhat MA. Laparoscopic management of adnexal abscesses: consequences for fertility. Fertil Steril. 1996 Nov;66(5):712-7. doi: 10.1016/s0015-0282(16)58623-3. PMID 8893672
- [Background] Heinonen PK, Leinonen M. Fecundity and morbidity following acute pelvic inflammatory disease treated with doxycycline and metronidazole. Arch Gynecol Obstet. 2003 Oct;268(4):284-8. doi: 10.1007/s00404-002-0376-6. Epub 2002 Oct 26. PMID 14504870
- [Background] Trent M, Bass D, Ness RB, Haggerty C. Recurrent PID, subsequent STI, and reproductive health outcomes: findings from the PID evaluation and clinical health (PEACH) study. Sex Transm Dis. 2011 Sep;38(9):879-81. doi: 10.1097/OLQ.0b013e31821f918c. PMID 21844746
- [Background] Ness RB, Soper DE, Holley RL, Peipert J, Randall H, Sweet RL, Sondheimer SJ, Hendrix SL, Amortegui A, Trucco G, Songer T, Lave JR, Hillier SL, Bass DC, Kelsey SF. Effectiveness of inpatient and outpatient treatment strategies for women with pelvic inflammatory disease: results from the Pelvic Inflammatory Disease Evaluation and Clinical Health (PEACH) Randomized Trial. Am J Obstet Gynecol. 2002 May;186(5):929-37. doi: 10.1067/mob.2002.121625. PMID 12015517
- [Background] Abbitt PL, Goldwag S, Urbanski S. Endovaginal sonography for guidance in draining pelvic fluid collections. AJR Am J Roentgenol. 1990 Apr;154(4):849-50. doi: 10.2214/ajr.154.4.2107687. No abstract available.
- [Background] Buchweitz O, Malik E, Kressin P, Meyhoefer-Malik A, Diedrich K. Laparoscopic management of tubo-ovarian abscesses: retrospective analysis of 60 cases. Surg Endosc. 2000 Oct;14(10):948-50. doi: 10.1007/s004640000249. PMID 11080409
- [Background] Henry-Suchet J, Soler A, Loffredo V. Laparoscopic treatment of tuboovarian abscesses. J Reprod Med. 1984 Aug;29(8):579-82. No abstract available. PMID 6237196
- [Background] Garbin O, Verdon R, Fauconnier A. [Treatment of the tubo-ovarian abscesses]. J Gynecol Obstet Biol Reprod (Paris). 2012 Dec;41(8):875-85. doi: 10.1016/j.jgyn.2012.09.012. Epub 2012 Nov 10. French. PMID 23146745
- [Background] Perez-Medina T, Huertas MA, Bajo JM. Early ultrasound-guided transvaginal drainage of tubo-ovarian abscesses: a randomized study. Ultrasound Obstet Gynecol. 1996 Jun;7(6):435-8. doi: 10.1046/j.1469-0705.1996.07060435.x. PMID 8807761
- [Background] Vermersch C, Dessein R, Lucot JP, Rubod C, Cosson M, Giraudet G. [Tubo-ovarian abscesses treatment: Faisability and results of trans-vaginal ultrasound-guided aspiration]. J Gynecol Obstet Biol Reprod (Paris). 2016 Mar;45(3):243-8. doi: 10.1016/j.jgyn.2015.04.016. Epub 2015 Jun 19. French. PMID 26096351